CLINICAL TRIAL: NCT06191757
Title: Effect Of Early Intervention Program Applied To Premature Infants In The Neonatal Intensive Care Unit On Comfort And Development
Brief Title: Effect Of Early Intervention Program Applied To Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, funda güler, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AydınAdnanMenderesUniversıty
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Infant Development; Patient Comfort; Nursing Caries; Premature Infant Disease
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The sample consisted of n=57 premature infants, n=27 in the study group and n=30 in the control group. Data were collected in two stages. In the first stage, mothers sang lullabies to the infants in the study group three times a week and touched them tenderly. In the second stage, developmental support program (GEDEP) was applied to the same infants for three months starting from the 40th week of gestation. The infants in the control group were given routine care. In data collection, Mother and Newborn Descriptive Information Form, Premature Infant Comfort Scale (PICS), Developmental Support Program Evaluation Form, GEDEP user guide form and Sound Decibel Measurement Device were used.
  Interventions: Behavioral: supported with the developmental support program
- control group (Experimental): The data of the control group were collected in two stages. No intervention was made to the control group by the researcher.
  First stage application steps:
  * Before starting the application, the Mother and Newborn Information Form (Annex 1) was filled out by the researcher.
  * The babies in the control group were cared for and their daily care (hygienic care (oral care, eye care, body care, diaper cleaning, etc.), feeding, taking vital signs, other follow-ups) were carried out by the nurse.
  Approximately 10-15 minutes and 20-25 minutes after the care was completed, the baby's responses were evaluated by the researcher with the premature comfort scale.
  Second stage: When the babies in the control group reached their first corrected month, developmental evaluations were made by the researcher using the GEDEP evaluation form every four weeks for a total of three months.
  Interventions: Behavioral: supported with the developmental support program

INTERVENTIONS:
Behavioral: supported with the developmental support program — Babies were developmentally supported with the developmental support program

SUMMARY:
Purpose: This study was conducted to evaluate the effect of singing a lullaby with compassionate touch on early comfort and later on development of developmental support program in premature infants in the neonatal intensive care unit.

H01: Singing a lullaby along with touching in the early stages of premature babies in the neonatal intensive care unit has no effect on the comfort score of the babies.

H02: Singing a lullaby along with touching to premature babies in the neonatal intensive care unit in the early period and then applying a developmental support program has no effect on the social emotional skills of premature babies.

H03: Singing lullabies with touch to premature babies in the neonatal intensive care unit in the early period and then applying a developmental support program has no effect on the language skills of premature babies.

H04: Singing a lullaby along with touching to premature babies in the neonatal intensive care unit in the early period and then applying a developmental support program has no effect on the cognitive skills of premature babies.

H05: Singing a lullaby along with touching to premature babies in the neonatal intensive care unit in the early period and then applying a developmental support program has no effect on the motor skills of premature babies.

DETAILED DESCRIPTION:
Materials and Methods: This study is a randomized controlled experimental study. The research was carried out in Aydın Adnan Menderes University Application and Research Hospital Neonatal Intensive Care Unit between 28 November 2021 and 18 July 2022. Premature infants at 330/7 -366/7 weeks of gestation who were hospitalized in the neonatal intensive care unit were included in the sampling. The sample consisted of n=57 premature infants, n=27 in the study group and n=30 in the control group. Data were collected in two stages. In the first stage, mothers sang lullabies to the infants in the study group three times a week and touched them tenderly. In the second stage, developmental support program (GEDEP) was applied to the same infants for three months starting from the 40th week of gestation. The infants in the control group were given routine care. In data collection, Mother and Newborn Descriptive Information Form, Premature Infant Comfort Scale (PICS), Developmental Support Program Evaluation Form, GEDEP user guide form and Sound Decibel Measurement Device were used. Data were evaluated with Chi-square test, Student's t-test and one-way analysis of variance, Mann-Whitney U test and Wilcoxon test. For repeated measurements, dependent groups t test and Wilcoxon signed-rank test were used.

ELIGIBILITY:
Inclusion Criteria:Criteria for including babies in the study;

* Premature babies born as singletons at 27-0/7 - 36-6/7 weeks of gestation,
* Premature babies whose corrected age was at the 40th week of gestation (to start the developmental support program)
* Mothers could speak, read and write Turkish were included in the study.

Exclusion Criteria:The exclusion criteria for babies from the study are as follows:

* Those diagnosed with perinatal or neonatal asphyxia, those with congenital anomalies, those with Stage 3-4 intracranial or intraventricular hemorrhage,
* Those who were given sedative opioids and anticonvulsant drugs
* Whose mothers had disabilities in communication (vision, hearing, speech)

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2021-11-28 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Premature Infant Comfort Scale (PICS), | on completion of the study ana average of 1 months
  PICS is a tool that multidimensionally evaluates the behavioral and psychological comfort and pain level of babies. In PBCS, Awakeness, Calmness/Agitation, Respiratory Status (only for those with mechanical ventilation support) or Crying (only for children with spontaneous breathing), Physical Movement, Muscle Tone, Facial Movements and Average Heart Rate are used to evaluate the baby's comfort level. Seven parameters are used. The scale is a 5-point Likert type scale where each parameter can be scored between 1 (bad) and 5 (good). According to PICS, the baby's comfort is evaluated based on the total score. The highest comfort score of 35 represents the lowest comfort score of 7. The total score determined as the cut-off value of the scale is 17. Babies with a total score of 17 or higher are considered cutoff for comfort level and indicate a need for pain-reducing interventions
GEDEP (Developmental Support Program) Evaluation Form | on completion of the study ana average of 3 months
  It aims to provide a rough assessment of children's cognitive, language/communication, motor, social-emotional and self-care skills in the 0-36 month period. This form contains introductory information such as the child's name, surname, date of birth, age, diagnosis, and parents' names. At the same time, skills in developmental areas included in GEDEP are also included in the form. Skills marked as "cannot do" and/or "partially able" on the form indicate the skills that the child needs to be worked on using GEDEP.

CONTACTS AND LOCATIONS:
Overall Officials: hüsniye çalışır, Prof, Study Director — study director
Locations (1):
- Funda Güler, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No